CLINICAL TRIAL: NCT02838901
Title: Dietary Nitrate Supplements and Ischemic Stroke Recovery: A Pilot Study
Brief Title: Dietary Nitrate Supplements and Ischemic Stroke Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00020739
Record Dates: First submitted 2016-06-19; First posted 2016-07-20 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Ischemic Stroke; Cerebrovascular Accident
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Beet It Beetroot Juice (Experimental): 70 cc (3.8 millimoles nitrate) Beet It organic beetroot juice once a day for 30 days. Vitamin C 500 mg (tablets) will be given along with each dose of the juice.
  Interventions: Drug: Beet it Beetroot juice
- Beet It Beetroot Juice Placebo (Placebo Comparator): 70 cc Beet It organic beetroot juice (placebo) once a day for 30 days. The placebo beet juice is identical in appearance and taste with nitrate removed. Vitamin C 500 mg (tablets) will be given along with each dose of the juice.Beet It Placebo Beetroot juice.
  Interventions: Drug: Beet It Placebo Beetroot juice

INTERVENTIONS:
Drug: Beet it Beetroot juice — Concentrated organic beetroot (98%) and lemon juice (2%); 70ml bottle
  Other Names: beetroot juice
  Arms: Beet It Beetroot Juice
Drug: Beet It Placebo Beetroot juice — Concentrated organic beetroot (98%) and lemon juice (2%) with nitrate extracted; 70ml bottle. Beet It Placebo Beetroot juice.
  Other Names: beetroot juice placebo
  Arms: Beet It Beetroot Juice Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, pilot study. Participants will be randomized to receive either beetroot juice or a beetroot juice placebo, as a dietary supplement, for 30 days. Beetroot juice is high in nitrates, a chemical when ingested is found to increase blood flow to the brain. The purpose of this research study is to determine the safety and feasibility of using this nutritional intervention in (ischemic)stroke survivors, and prove that plasma levels of nitrate and nitrite increase as expected. Secondary outcomes includes measuring a comprehensive set of outcomes related to functional status post-stroke, including mobility, upper extremity strength, cognition, depression, and disability. Patients will also be randomized to MRI perfusion scanning in the region of the stroke to measure cerebral blood flow.

DETAILED DESCRIPTION:
In this proof of concept study, the investigators will for the first time, determine whether dietary nitrate (commercially available beetroot juice) is safe and feasible to administer in ischemic stroke patients, and whether its use is associated with increased plasma nitrate and nitrite levels and trends toward improvement during the standard 30-day rehabilitation period after a stroke. The investigators will test the hypotheses using a double-blinded randomized placebo-controlled trial of Beet It® shots once daily for 30 days for patients enrolled within 5 days of stroke onset. This novel study will provide key safety and feasibility data on dietary nitrate supplementation and preliminary information on the magnitude of its effect on improving mobility and functional status, cognition and cerebral blood flow. These data are needed to accelerate the pace of development of this novel therapeutic strategy: using a non-pharmacological approach for improving stroke outcomes. The specific aims are to: Aim 1) Test the proof of concept that beetroot juice consumption is feasible and safe in ischemic stroke patients when given during the post-acute rehabilitation period. Primary outcomes are adherence to the intervention, measurement of outcomes and follow-up (feasibility), as well as adverse events (safety), reported as proportions in each group and across the entire study cohort. Hypothesis: Beetroot juice is safe and feasible in this population, and leads to increased plasma nitrate and nitrite levels at 30 days. Secondary outcomes of interest include change in gait speed (m/sec), Modified Rankin score (disability scale), NIHSS, EuroQOL-5D (quality of life),Patient Health Questionnaire-9 (depression), Stroke Impact Scale-16 (SIS-16), Barthel Index, Short Physical Performance Battery, grip strength and the Montreal Cognitive Assessment (MoCA). Aim 2) Determine whether beetroot juice consumption increases cerebral blood flow vs. placebo juice. Cerebral blood flow will be determined from MRI collected 2 hours following ingestion of the beetroot juice on day 30. Anatomic and perfusion imaging (PASL) will be performed. A region of interest will be used to measure blood flow in a 20mm sphere placed adjacent to the ischemic stroke and in the contralateral hemisphere. Hypothesis: Ischemic stroke patients randomized to the beetroot juice intervention will show increased cerebral blood flow as measured by MRI perfusion scanning in the region of the stroke compared with the placebo group at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and over
* Diagnosed with an ischemic stroke (acute focal neurological deficit resulting from an ischemic cause, verified by CT or MRI)
* Symptom onset within 5 days of admission
* National Institutes of Health Stroke Scale Score of 2 or more (but less than 20)
* A rating of fair or good on static sitting balance scale on a global balance scale
* A score of more that 0 on the hip flexion on the short Fugl-Myer
* Passed dysphagia screening for unrestricted or thickened liquids

Exclusion Criteria:

* Patients with severe stroke (National Institutes of Health Stroke Scale Score of 20 or more)
* A score of 0 on hip flexion on the Short Fugl-Myer as a result of weakness from the stroke
* A rating of poor on static sitting balance scale on a global balance scale
* Patients who received intravenous or intra-arterial recombinant tissue plasminogen activator (rtPA)
* Patients who are receiving citicoline
* Patients who have had a hemorrhagic stroke (including intraparenchymal, subarachnoid or subdural hemorrhage)
* A gait speed of more > 0.8 m/s
* Patient with evidence of brain tumor or other psychiatric or neurological condition that would interfere with outcome measures
* Patients who will undergo carotid endarterectomy or other surgery during the study period
* Patients not living independently prior to stroke
* Survival is expected to be less than 6 months
* Any patient on organic nitrate-containing medications; some examples of the medications that are exclusions include nitroglycerin, isosorbide mononitrate, sildenafil (Viagra), and tadalafil (Cialis)
* Patients with atrophic gastritis
* Patients with hypotension (blood pressure less than 100/60 mmHg)
* Patients who do not pass the dysphagia screening test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Bushnell, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will be notified as to which arm of the study they were randomized to. The de-identified participant data will be presented as an abstract, if accepted, and published as a manuscript.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled adults who have suffered an ischemic stroke with minimum impairments defined by NIHSS scores and physical function measurements.
Pre-assignment Details: From June 2012 to June 2016, patients who are admitted to the Stroke Unit and who are within 96 hours of symptom onset, were screened for eligibility by reviewing their admitting history and physicals and imaging results.
Groups:
- Beet It Beetroot Juice: 70 cc (3.8 millimoles nitrate) Beet It organic beetroot juice once a day for 30 days. Vitamin C 500 mg (tablets) will be given along with each dose of the juice.
  Beet it Beetroot juice: Concentrated organic beetroot (98%) and lemon juice (2%); 70ml bottle.
  Nine participants were randomized to the Beet It Beetroot Juice arm. Participants had blood drawn on study day 1 and day 30 for nitrate and nitrite levels before and one hour after drinking 70 cc (3.8 mM nitrate) plus vitamin C 500 mg daily. On day 30, gait speed (using the 4 m walk) was assessed.
  Eighteen participants were consented, 15 completed treatment (1 terminated treatment because of nausea), 16 followed for 30 days and 13 for 90 days.
  Participants selected for the MRI portion of the study had a brain MRI performed on study day 30 to measure cerebral blood flow.
- Beet It Beetroot Juice Placebo: 70 cc Beet It organic beetroot juice (placebo) once a day for 30 days. The placebo beet juice is identical in appearance and taste with nitrate removed. Vitamin C 500 mg (tablets) will be given along with each dose of the juice.Beet It Placebo Beetroot juice.
  Beet It Placebo Beetroot juice: Concentrated organic beetroot (98%) and lemon juice (2%) with nitrate extracted; 70ml bottle. Beet It Placebo Beetroot juice.
  Nine participants were randomized to the Beet It Beetroot Juice Placebo arm. Participants had blood drawn on study day 1 and day 30 for nitrate and nitrite levels before and one hour after drinking 70 cc (3.8 mM nitrate) plus vitamin C 500 mg daily. On day 30, gait speed (using the 4 m walk) was assessed.
  Eighteen participants were consented, 15 completed treatment (1 terminated treatment because of nausea), 16 followed for 30 days and 13 for 90 days.
  Participants selected for the MRI portion of the study had a brain MRI performed on study day 30 to measure cerebral b
Period: Overall Study
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Started | 9 | 9
Completed | 7 | 7
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were balanced with regard to admission NIHSS, age, sex, race, risk factors, baseline gait speed, and baseline nitrate/nitrite levels.
Groups:
- Total: Total of all reporting groups
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Age (yrs)] | 63.5 (8.6) | 66.3 (9.2) | 64.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 5 | 7 | 12
  More than one race | NA — more than one race reported as other/unknown | NA — more than one race reported as other/unknown | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18
nitrate and nitrite levels [Mean (Standard Deviation); unit: micromoles/L]
  Baseline Nitrate | 63.9 (77.2) | 27.0 (16.0) | 45.5 (57.3)
  Baseline Nitrite | 0.17 (0.14) | 0.13 (0.08) | 0.15 (0.11)
gait speed [Mean (Full Range); unit: m/s] — Population: A total of 17 participants had baseline gait speed data available
  m/s
    number analyzed (Participants) | 8 | 9 | 17
    (all) | 0.23 [0.07 to 0.36] | 0.22 [0.08 to 0.23] | 0.22 [0.08 to 0.32]

OUTCOME MEASURES:

1. Primary Outcome: Adherence With Intervention
Description: The primary outcome for this trial is feasibility, which will be measured by how well the participants followed instructions on taking Beet It organic beetroot juice or placebo once a day for 30 days.
Time Frame: 30 days
Population: Two participants were lost to follow-up by 30 days, therefore the analysis included 8 participants in each group.
Measure: Mean (Inter-Quartile Range); unit: percentage of participants
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 8 | 8
percentage of participants | 93.5 [80 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; The null hypothesis was used, and the assumption was there would be no difference in adherence between the Active Juice and the Placebo Juice, and therefore a two-sided t approximation was reported. Since this was a pilot study, power calculations were not performed. The adherence in the two groups was compared using the Wilcoxon two-sample test; Test type: Other — This was a descriptive analysis, and was based on the overall assessment of feasibility of the intervention; p = 0.058, Wilcoxon (Mann-Whitney) — The p value is not adjusted for multiple comparisons

2. Primary Outcome: Number of Participants With Adverse Treatment-altering Events
Description: Adverse events that lead to treatment discontinuation
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 9 | 9
participants | 1 | 0
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Null hypothesis was assumed, no power calculation was done since this was a pilot study; Test type: Other — This was a descriptive analysis and was under the goal of assessing safety of the intervention; p = 1.00, Fisher Exact

3. Primary Outcome: Change in Plasma Nitrate Levels, Micromoles/Liter
Description: This is the proof-of-concept to see if plasma levels change in those randomized to the active beet juice compared to placebo. Comparing baseline values against values at 30 days.
Time Frame: after 30 days of treatment
Population: The median treatment-specific changes in nitrate were analyzed using comparison of pre to post-dosing plasma on day 1. Beetroot It Beetroot juice (Active) was associated with an increase in plasma nitrate and a trend towards increased nitrite levels. The analysis included 8 participants per group since 2 did not come back for follow-up at 30 days.
Measure: Median (Inter-Quartile Range); unit: micromoles/L
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 8 | 7
micromoles/L | 174.76 [149.68 to 241.09] | 0.678 [-1.678 to 2.060]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; The null hypothesis was assumed, and no power calculation was performed since this was a pilot study; Test type: Other; p = 0.0003, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Plasma Nitrite Levels, Micromoles/Liter
Description: as for outcome 3
Time Frame: after 30 days of treatment
Population: The median treatment-specific changes in nitrate were analyzed using comparison of pre to post-dosing plasma on day 1. Beetroot It Beetroot juice (Active) was associated with an increase in plasma nitrate and a trend towards increased nitrite levels. The analysis included 8 participants in active and 7 in placebo based on follow-up at 30 d.
Measure: Median (Inter-Quartile Range); unit: micromoles/L
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 8 | 7
micromoles/L | 0.114 [0.044 to 0.158] | 0.014 [0.002 to 0.028]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other — This was a descriptive analysis for a pilot study, and no power calculations were performed; p = 0.1023, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Gait Speed Change From Baseline
Description: Gait speed is measured by the time it takes to walk 10 meters. Baseline was reported.Change in gait speed from baseline was assessed at 30 and 90 days. Non-ambulatory at baseline is defined as gait speed less than 0.1 m/s.
Time Frame: baseline, 30, and 90 days
Population: There were 8 participants in the Active and 8 in the placebo because they did not follow-up at 30 days. BL ambulatory refers to only those participants were able to walk at baseline immediately after enrollment. For this analysis, there were only 6 participants in the active and 7 in the placebo at 30 days and 4 and 5 at 90 days, respectively.
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 8 | 8
m/s
  Baseline | .22 [.08 to .32] | .23 [.07 to .36]
  Gait speed change 30 days | 0.330 [0.049 to 0.498] | 0.193 [0.000 to 0.590]
  Gait speed change 90 days | 0.385 [0.030 to 0.635] | 0.165 [0.000 to 0.760]
  BL Ambulatory: Gait Speed 30 days: number analyzed (Participants) | 6 | 7
  BL Ambulatory: Gait Speed 30 days | 0.591 [0.180 to 0.910] | 0.575 [0.326 to 1.060]
  BL Ambulatory: Gait Speed 90 days: number analyzed (Participants) | 4 | 5
  BL Ambulatory: Gait Speed 90 days | 0.572 [0.275 to 0.942] | 0.406 [0.240 to 1.220]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other — This was a descriptive analysis for a pilot study to gather preliminary data for a larger trial. No power calculations were performed for this outcome; p = .9581, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; The null hypothesis was assumed, and no power calculation was performed since this was a pilot study and the purpose was to collect preliminary data for a larger trial; Test type: Other; p = .6678, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Cerebral Perfusion Imaging
Description: Participants from each group who had an MRI at baseline will be randomly selected to have a repeat MRI perfusion scan at 30 days. Cerebral blood flow will be measured by MRI perfusion scanning (arterial spin labeling) in the region of the stroke.
Time Frame: 30 days
Population: MRI cerebral perfusion data could not be analyzed because of a change in the measurement of perfusion after the first participant was enrolled.
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Upper Extremity Grip Strength
Description: The hand grip strength test is designed to replicate the grip strength required to undertake officer survival and firearms training. The test is completed using a dynamometer which measures grip strength in kilograms (kg). The score ranges from 0-90kg, higher score denotes better outcomes.
Time Frame: 30 days
Population: Only 6 participants in each group had grip strength measured at 30 days. Affected refers to the upper extremity that was affected by the stroke, and unaffected refers to the upper extremity not affected by the stroke.
Measure: Mean (Inter-Quartile Range); unit: kg
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 6 | 6
kg
  Affected | 17.4 [11.5 to 32.5] | 20 [11 to 35]
  Unaffected | 28.75 [22 to 49.4] | 34.75 [21.5 to 38.7]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = .876, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Upper Extremity Grip Strength
Description: The hand grip strength test is designed to replicate the grip strength required to undertake officer survival and firearms training. The test is completed using a dynamometer which measures grip strength in kilograms. The score ranges from 0-90kg, higher score denotes better outcomes.
Time Frame: 90 days
Population: Only 6 in the active and 7 in the placebo had grip strength measured at 90 days. Affected refers to the upper extremity that was affected by the stroke, and unaffected refers to the upper extremity not affected by the stroke.
Measure: Mean (Inter-Quartile Range); unit: kg
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 6 | 7
kg
  Affected | 17.5 [8 to 22.7] | 11 [3 to 27]
  Unaffected | 26.75 [19.5 to 31.3] | 33 [23 to 85]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = .889, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = 0.532, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Montreal Cognitive Assessment (MoCA) Score
Description: Cognition is measured with the Montreal Cognitive Assessment. MoCA is a 30 question test that assesses different types of cognitive abilities, including orientation, short-term memory, executive function, language abilities, attention and visuospatial ability. Scores on the MoCA range from zero to 30, higher scores denotes better outcomes.
Time Frame: 30 days
Population: Only 5 participants in the active and 8 in the placebo were able to complete the MoCA at 30 days.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 5 | 8
units on a scale | 23.5 [19 to 27] | 23 [20 to 25]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = 0.888, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Montreal Cognitive Assessment (MoCA) Score
Description: Cognition is measured with the Montreal Cognitive Assessment. Cognition is measured with the Montreal Cognitive Assessment. MoCA is a 30 question test that assesses different types of cognitive abilities, including orientation, short-term memory, executive function, language abilities, attention and visuospatial ability. Scores on the MoCA range from zero to 30, higher scores denotes better outcomes.
Time Frame: 90 days
Population: Only 5 participants in the active and 8 in the placebo were able to complete the MoCA at 90 days.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 5 | 8
units on a scale | 27 [24 to 29] | 23.5 [19.5 to 26.5]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = 0.475, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Modified Rankin Score
Description: Modified Rankin Scale is a measure of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scores range from 0 (no symptoms) to 5 (bedridden in a nursing home). Lower scores denotes better outcomes.
Time Frame: 30 days
Population: Only 8 participants in the active and 8 in the placebo returned for the 30 day visit in order to measure the modified Rankin score.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 8 | 8
units on a scale | 3 [1 to 3] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = 0.135, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Modified Rankin Score
Description: as for outcome 11
Time Frame: 90 days
Population: Only 6 participants in the active and 8 in the placebo returned for the 90 day visit and therefore modified Rankin could not be ascertained.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
Number analyzed (Participants) | 6 | 8
units on a scale | 2.5 [1 to 3] | 3 [2.5 to 5]
Statistical Analysis 1: Comparison: Beet It Beetroot Juice vs Beet It Beetroot Juice Placebo; Test type: Other; p = 0.185, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Beet It Beetroot Juice | Beet It Beetroot Juice Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/9 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beet It Beetroot Juice (N=9) | Beet It Beetroot Juice Placebo (N=9)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Beet It Beetroot Juice (N=9) | Beet It Beetroot Juice Placebo (N=9)
Stroke (Nervous system disorders) | 1 (1) | 1/1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastroesophageal refluix (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Easy bruising (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Mental alteration (Nervous system disorders) | 1 (1) | 0 (0)
Hypothermia (Endocrine disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Hyperkalemia (Endocrine disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chest Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Non-specific SA nodal disease (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (General disorders) | 0 (0) | 1 (2)
Eye floater (Eye disorders) | 0 (0) | 1 (2)
Fall (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No